CLINICAL TRIAL: NCT00991120
Title: Extension Phase of the Chronicle® Offers Management to Patients With Advanced Signs & Symptoms of Heart Failure Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: COMPASS-HF Extension
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Chronicle Implantable Hemodynamic Monitor (IHM) System, Chronicle Implantable Cardioverter Defibrillator (ICD) — Surgical implantation of chronic ambulatory hemodynamic monitoring device and intracardiac lead
  Other Names: Chronicle IHM, Chronicle ICD

SUMMARY:
The purpose of the Extension Phase of the COMPASS-HF study is to continue to observe the safety of the Chronicle® Implantable Hemodynamic Monitor (IHM) system and Chronicle ICD system and provide study doctors continued access to the heart pressure information recorded by the Chronicle devices which may be used to help manage heart failure. The Extension Phase of the COMPASS-HF study is limited to people who have already received the investigational system and are currently enrolled in a Chronicle IHM or ICD study.

DETAILED DESCRIPTION:
For the purpose of the Extension Phase, the Chronicle IHM and ICD systems are for continued use in patients with moderate to severe heart failure and are intended to monitor hemodynamic information, including right ventricular and pulmonary artery pressures, heart rate and activity. The COMPASS-HF Extension Phase includes the following Chronicle IHM studies:

* The Chronicle IHM Phase I/II study, which was a 148 patient technology assessment study that began enrolling patients in 1998 and completed the endpoint driven follow up period of 3 months for safety and 12 months for efficacy in 2002
* The Chronicle Offers Management to Patients with Advanced Signs & Symptoms of Heart Failure (COMPASS-HF) study, which was a 274 patient randomized study that began enrolling patients in 2003 and completed the endpoint driven follow up period of 6 months in 2005
* The Pulmonary Arterial Hypertension Pilot (PAH Pilot) study, which was a 24 patient pilot study that began enrolling patients in 2003 and completed the endpoint driven follow up period of 12 weeks in 2006
* The Reducing Decompensation Events Utilizing intraCardiac Pressures in Patients with Chronic HF (REDUCEhf) study, which was a 400 patient randomized study that began enrolling patients in 2006 and completed endpoint driven follow up period of 12 months in 2010.

In all four studies, patients were implanted with a Chronicle IHM or ICD system and upon completion of the endpoint driven follow up period, entered long term follow up and have continued to be seen every six months for study visits.

As the Chronicle IHM or ICD system has not received U.S. Food and Drug Administration approval, the COMPASS-HF Extension Phase is being initiated as a means to allow continued access of Chronicle IHM data to study investigators in one concurrently enrolled study and follow up schedule. No additional study objectives or new enrollments will be captured in the COMPASS-HF Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides written informed consent for the Extension Phase
* Patient has an implanted Chronicle IHM or ICD device and is actively enrolled in one of the following studies: COMPASS-HF, Chronicle IHM Phase I/II, REDUCEhf or the PAH Pilot Study

Exclusion Criteria:

* Patient unwilling to transmit their Chronicle IHM or ICD device data as directed by their study clinicians or unwilling to participate in protocol scheduled follow up visits (every six months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all currently enrolled patients in the COMPASS-HF, Chronicle IHM Phase I/II, REDUCEhf and PAH Pilot studies who provide written informed consent for the Extension Phase.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COMPASS-HF Extension Team, Study Chair — Medtronic
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Davenport, Iowa
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - New Brunswick, New Jersey
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia